CLINICAL TRIAL: NCT06084052
Title: Path Active Multicentre Randomised Controlled Trial (Previous Pilot: Path Active; Safety and Tolerability Study)
Acronym: PAMRCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Free Hospital NHS Foundation Trust (Other)
Collaborators: Walk With Path (Industry)
Responsible Party: Principal Investigator, Richard Leigh, Chief Investigator, Royal Free Hospital NHS Foundation Trust
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 326601
Record Dates: First submitted 2023-08-22; First posted 2023-10-16 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Diabetic Foot
Keywords: Foot Ulcer Prevention
MeSH Terms: conditions — Diabetic Foot | interventions — Control Groups

STUDY DESIGN:
Masking Description: The participants will be randomised (using 'sealed envelope') to either 'care as usual' or 'use of device'.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Path Active (Other): Participants randomised to use the device
  Interventions: Device: Path Active
- Control Group (Other): Participants randomised to care as usual
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Path Active — Participant use of Path Active insoles, mobile phone app and clinician's dashboard (where pressure and temperature changes can be reviewed by a clinician). All participants will complete a patient questionnaire relating to use of the device and EuroQol - EQ5D at the beginning and end of the study.
  Arms: Path Active
Other: Control Group — Control Group will receive care as usual.
  Arms: Control Group

SUMMARY:
Path Active™ comprises a pair of monitoring insoles which measure parameters associated with foot ulceration in diabetes: temperature and pressure. The insoles are linked via an app to the wearer's mobile phone and also to a clinical dashboard so that both wearer and clinician are alerted to early signs of skin damage on the foot so that immediate preventive action can be taken. The study is a multisite randomised controlled trial which will evaluate the effectiveness of Path Active™ in 60 people with diabetes who are at 'high risk' of foot ulceration, compared with 60 people who receive their usual podiatry foot checks over a period of 12 weeks.

DETAILED DESCRIPTION:
Foot complications in people with diabetes are the most common cause of non-traumatic leg amputation in the UK with over 176 leg, toe or foot amputations every week in England. One in seven people with diabetes will develop a foot ulcer at some stage in their lives. Not only does this impair their daily activities and reduce their quality of life, it also increases their risk of amputation by up to 24-fold. Five year mortality for minor and major amputations in diabetes have been reported as 46.2% and 56.6%, respectively. Circulatory problems, nerve impairment and infection contribute to foot complications in diabetes. Prior to a foot ulceration, changes in temperature and/or pressure occur. These early warning signs can be measured by Path Active™ and alert the wearer via a mobile phone app and the clinician via a clinical dashboard so that preventive action can be taken. Currently people with diabetes who have been assessed as 'high risk' for foot ulceration are allocated appointments with podiatrists in 'foot protection teams' who review on a weekly to monthly basis. Path Active™ has the potential to reduce appointments by alerting podiatry teams to potential problems as they occur rather than regular routine reviews. Path Active™ may be able to reduce hospital and clinic visits and thereby reduce healthcare carbon footprint.

The primary objective of this clinical investigation is to evaluate the effectiveness of Path Active™ in people with diabetes who are at 'high risk' of foot ulceration. The study is a multisite randomised controlled trial which will evaluate the effectiveness of Path Active™ in 60 people with diabetes who are at 'high risk' of foot ulceration, compared with 60 people who receive their usual podiatry foot checks over a period of 12 weeks. Recruitment to the study will be in 4 clinical sites across England and Scotland.

The protocol for this study was amended from the pilot study and accepted as a 'major amendment' by the regional Ethics Committee of Essex. Therefore the IRAS number (Unique Protocol ID: 326601) has remained the same.

ELIGIBILITY:
Inclusion Criteria:

* • Participant able to give informed consent.
* Age >18 at the time of consent.
* Diagnosis of Type 1 or Type 2 Diabetes.
* Both Feet Intact (no ulceration).
* Participant understands and is willing to participate and can comply with the follow-up regime.
* Participant diabetes foot Risk Stratification as 'High Risk' as in Frame (2021) Scotland/England https://www.diabetesframe.org/
* Ability to walk independently for > 100 metres i.e without use of wheelchair, walking stick or personal assistance.
* Participant able and willing to wear suitable footwear.
* Must own a mobile phone and be willing to upload WWP app.

Exclusion Criteria:

* Either foot has less than 2 arterial vessel run-off on Doppler.
* Poor visual acuity ie registered blind, unless supported by carer.
* Current participation in another clinical investigation of a medical device or a drug; or participation in such a study within 30 days prior to study enrolment.
* Body Mass Index (BMI) >40.
* Participant has bespoke contact insoles and footwear.
* Participant is unable to use 'medium' or 'large' insoles due to foot size eg. small or extra large feet.
* Participant has a pacemaker.
* Participant is pregnant.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 months (Participants will wear the device for a minimum of 7 days)
  The primary objective of this clinical investigation is to evaluate the effectiveness of Path Active™ in people with diabetes who are at 'high risk' of foot ulceration.
Changes Quality of Life Measurement | 6 months (Participants will wear the device for a minimum of 12 weeks)
  EuroQol EQ-5D-5L assessment for quality of life assessment at the beginning and end of the study period.
  The EQ-5D-5L health profile includes the items mobility (MO), self-care (SC), usual activities (UA), pain/discomfort (PD) and anxiety/depression (AD). The EQ-5D-5L asks respondents to endorse one of five response levels for each item: "no problems," "slight problems," "moderate problems," "severe problems," and "extreme problems"/ "unable to", describing 3125 (55) health state profiles. The instrument also includes a visual analog scale (VAS) anchored by 0 (worst imaginable health) and 100 (best imaginable health) that will be analysed separately from the health profile.
Device questionnaire | 6 months (Participants will wear the device for a minimum of 12 weeks)
  Participants in the 'Path Active' arm will complete study questionnaires relating to the product (ease of use, use of the mobile phone app, use of the insoles, action taken relating to app warnings).
Control Group questionnaire | 6 months
  Participants in the 'Control Group' arm will complete study questionnaires relating to their usual care (how often do you see a healthcare professional for foot checks, how often do you examine your feet, how concerned are you about developing a foot ulcer etc)

SECONDARY OUTCOMES:
Reduction in CO2 comparing carbon dioxide emitted due to ulcer treatment vs carbon dioxide emitted due to device manufacture | 6 months (Participants will wear the device for a minimum of 12 weeks)
  To model the carbon dioxide reduction that occurs if ulceration and the need for ulcer treatment is prevented, in differing UK geographies. The carbon footprint for the manufacture and life span of the device will been calculated and the carbon footprint for ulcer treatment will be calculated. The difference between CO2 due to manufacture of the device will be compared with the CO2 required for ulcer treatment to show how much reduction in carbon can be made by preventing foot ulceration when using Path Active.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Leigh, BSc, Study Chair — Royal Free London NHS Foundation Trust
Locations (1):
- Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbott CA, Chatwin KE, Foden P, Hasan AN, Sange C, Rajbhandari SM, Reddy PN, Vileikyte L, Bowling FL, Boulton AJM, Reeves ND. Innovative intelligent insole system reduces diabetic foot ulcer recurrence at plantar sites: a prospective, randomised, proof-of-concept study. Lancet Digit Health. 2019 Oct;1(6):e308-e318. doi: 10.1016/S2589-7500(19)30128-1. Epub 2019 Sep 26. PMID 33323253
- [Result] Armstrong DG, Boulton AJM, Bus SA. Diabetic Foot Ulcers and Their Recurrence. N Engl J Med. 2017 Jun 15;376(24):2367-2375. doi: 10.1056/NEJMra1615439. No abstract available. PMID 28614678
- [Result] Chatwin KE, Abbott CA, Boulton AJM, Bowling FL, Reeves ND. The role of foot pressure measurement in the prediction and prevention of diabetic foot ulceration-A comprehensive review. Diabetes Metab Res Rev. 2020 May;36(4):e3258. doi: 10.1002/dmrr.3258. Epub 2019 Dec 11. PMID 31825163
- [Result] Kerr M, Barron E, Chadwick P, Evans T, Kong WM, Rayman G, Sutton-Smith M, Todd G, Young B, Jeffcoate WJ. The cost of diabetic foot ulcers and amputations to the National Health Service in England. Diabet Med. 2019 Aug;36(8):995-1002. doi: 10.1111/dme.13973. Epub 2019 Jun 5. PMID 31004370

DOCUMENTS (2):
  • Study Protocol (2024-06-12): https://cdn.clinicaltrials.gov/large-docs/52/NCT06084052/Prot_002.pdf
  • Informed Consent Form (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT06084052/ICF_003.pdf